CLINICAL TRIAL: NCT03948022
Title: Which Luteal Support in Frozen-Thawed Embryo Transfer Cycles: A Randomized Controlled Trial
Brief Title: Luteal Support in Frozen-Thawed Embryo Transfer Cycles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centrum Clinic IVF Center (Other)
Responsible Party: Principal Investigator, Emre Göksan Pabuçcu, Associated Professor, Centrum Clinic IVF Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: centrumtupbebek
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Implantation; Placenta; Pregnancy Loss; Frozen Embryo; Luteal Support; Luteal Phase Defect; Assisted Reproduction
Keywords: progesterone; implantation; pregnancy; abortion
MeSH Terms: interventions — Dydrogesterone; Tablets; Progesterone; Oils; Crinone; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intramuscular progesterone (Active Comparator): progestan (progesterone) 50 mg/ml ampoules, 2 ampoules (100 mg) intramuscular starting from day 11 of the endometrial preparation cycle.
  Interventions: Drug: Progesterone 50Mg/mL Oil
- vaginal progesterone (Active Comparator): crinone %8 bioadhesive gel (progesterone) 90 mg, twice daily (180 mg/day) starting from day 11 of the endometrial preparation cycle.
  Interventions: Drug: Crinone 8% Vaginal Gel
- oral dydrogesterone (Experimental): oral dydrogesterone (progesterone) 10 mg tablets, 2x2 (40 mg total)
  Interventions: Drug: Dydrogesterone 10Mg Tablet (duphaston)

INTERVENTIONS:
Drug: Dydrogesterone 10Mg Tablet (duphaston) — 40 mg daily oral tablets
  Arms: oral dydrogesterone
Drug: Progesterone 50Mg/mL Oil — 100 mg daily intramuscular injections
  Arms: intramuscular progesterone
Drug: Crinone 8% Vaginal Gel — 180 mg daily vaginal gels
  Arms: vaginal progesterone

SUMMARY:
This study evaluates the clinical efficacy of 3 different luteal phase support in patients undergoing frozen-thawed embryo transfer cycles. Endometrium preparation will be hormone replacement in all cycles. Starting from day 11, group 1 will receive 100 mg micronized progesterone parenteral daily injections, group 2 will receive 90 mg bioadhesive gel vaginal twice daily and group 3 will receive 40 mg oral dydrogesterone daily tablets.

DETAILED DESCRIPTION:
In natural pregnancy, successful implantation and pregnancy necessitates well-functioning corpus luteum. Luteal phase support (LPS) is critical in assisted conception cycles particularly for replacement frozen embryo transfer cycles owing to lack of corpus luteum. 3 different LPS options have been suggested:

* Progesterone in oil (intramuscular injections) is rapidly absorbed after i.m. injection and high progesterone plasma concentrations are reached after approximately 2h. Despite satisfactory plasma levels, the possible side-effects of pain and swelling are limiting the use.
* Vaginal application of progesterone is widely accepted with satisfactory endometrial levels and patient convenience. However, increased vaginal discharge and possible vaginal irritation are the most common side effects.
* Oral administration of synthetic progesterone (dydrogesterone) would offer a convenient way of progesterone administration. Better bioavailability than natural progesterone and less cost makes dydrogesterone preferable. Also, good quality evidence revealed satisfactory outcomes in fresh embryo transfer cycles. However, there is lack of good quality evidence for dydrogesterone as a LPS in frozen-thawed cycles.

The investigator's aim is to compare 3 widely used LPS in frozen-thawed embryo transfer cycles.

Following allocation of the subjects, hormone replacement will be scheduled for the endometrial preparation. Briefly; On day 2 of menstrual bleeding, endometrial preparation with oral estradiol (E2) (2 mg twice daily) will be initiated. Approximately 10 days after initiation of E2 administration, the subject will undergo a transvaginal ultrasound examination to assess endometrial development and serum progesterone (P) level will be checked. Once the subject achieved a trilaminar endometrium with a thickness of >7 mm with serum P levels <1.5 ng/ml, she will start the progesterone treatment to which she will be randomized to one of the 3 arms. After 3 days of P treatment along with E2 pills, cleavage embryo transfer will be performed. If the subject will receive blastocyst, 5 days of P treatment will be scheduled.

If these criteria were not met at the first evaluation, she will allowed up to 10 additional days (20 days total) of estrogen stimulation.

ELIGIBILITY:
Inclusion Criteria:

* woman aged 20-40 years
* Having available blastocyst(s) cryopreserved by vitrification method.

Exclusion Criteria:

* requirement for fresh embryo(s);
* presence of any clinically relevant systemic disease contraindicated for assisted reproduction or pregnancy
* history of more than three failed cycles of IVF
* history of recurrent abortions
* allergy history for relevant drugs
* body mass index of <18 or >38 kg/m2 at screening
* current breastfeeding or pregnancy
* refusal or inability to comply with the requirements of the protocol for any reason, including scheduled clinic visits and laboratory tests
* trophectoderm or blastomere biopsy of the blastocyst(s) to be transferred

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate | 12th week of pregnancy
  fetal cardiac activity beyond 12th week of gestation

SECONDARY OUTCOMES:
clinical pregnancy rate | 6th week of pregnancy
  fetal cardiac activity
abortion rate | during first 10 weeks of gestation
  miscarriage of the pregnancy pregnancy recently confirmed with positive beta hCG blood test

CONTACTS AND LOCATIONS:
Overall Officials: Emre Pabuccu, Assoc. Prof., Study Director — Ufuk University School of Medicine
Locations (1):
- Ufuk University School of Medicine, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Devine K, Richter KS, Widra EA, McKeeby JL. Vitrified blastocyst transfer cycles with the use of only vaginal progesterone replacement with Endometrin have inferior ongoing pregnancy rates: results from the planned interim analysis of a three-arm randomized controlled noninferiority trial. Fertil Steril. 2018 Feb;109(2):266-275. doi: 10.1016/j.fertnstert.2017.11.004. Epub 2018 Jan 17. PMID 29338855
- [Result] Griesinger G, Blockeel C, Sukhikh GT, Patki A, Dhorepatil B, Yang DZ, Chen ZJ, Kahler E, Pexman-Fieth C, Tournaye H. Oral dydrogesterone versus intravaginal micronized progesterone gel for luteal phase support in IVF: a randomized clinical trial. Hum Reprod. 2018 Dec 1;33(12):2212-2221. doi: 10.1093/humrep/dey306. PMID 30304457
- [Result] Zarei A, Sohail P, Parsanezhad ME, Alborzi S, Samsami A, Azizi M. Comparison of four protocols for luteal phase support in frozen-thawed Embryo transfer cycles: a randomized clinical trial. Arch Gynecol Obstet. 2017 Jan;295(1):239-246. doi: 10.1007/s00404-016-4217-4. Epub 2016 Oct 19. PMID 27761732